CLINICAL TRIAL: NCT01396473
Title: Study on Out of School Nutrition and Physical Activity Environments
Acronym: OSNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Steven Gortmaker/Professor of the Practice of Health Sociology, Department of Society, Human Development and Health; Harvard School of Public Helath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18046; CDC Grant Number (Other Grant/Funding Number: Centers for Disease Control and Prevention/1 -U48-DP-001946)
Record Dates: First submitted 2011-01-27; First posted 2011-07-18 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Child Physical Activity; Child Nutrition
Keywords: afterschool; accelerometers; plate waste; policy; environment
MeSH Terms: interventions — Policy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention)
- Policy and Environmental Change (Experimental)
  Interventions: Behavioral: Policy and Environmental Change

INTERVENTIONS:
Behavioral: Policy and Environmental Change — Afterschool programs participate in an assessment of physical activity and nutrition practices and policies. Study staff work with teams of afterschool programs in a participatory manner to identify areas in which programs would like to take practice, policy and communication efforts to meet physical activity and nutrition goals. Teams share progress and barriers during ongoing collaborative meetings.
  Arms: Policy and Environmental Change

SUMMARY:
The purpose of this study is to design and conduct research to tailor out of school time evaluation materials so they are applicable to various settings in Boston, are efficient in that minimal resources and time are used, and are useful to participants.

DETAILED DESCRIPTION:
Nearly half of Boston's school age children (49%) participate in out of school time programs, a critical time to intervene on physical activity and nutrition. Previous research has mostly focused on during-school-day efforts, or on child care policies and practices for very young children, leaving a gap in the knowledge of what might work with programs serving school-age children during out of school time. OSNAP aims to implement low cost and sustainable policy and environmental interventions to improve physical activity and healthy eating/beverage environments. Data will be collected via observations, plate waste and accelerometers on program policies, environments, practices and behavioral outcomes related to physical activity, beverage, snack and screen time outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Afterschool programs in Boston MA serving at least 40 children ages 5-12 years operating the full school year between September and June
* Afterschool programs serving a snack to children
* Children between the ages of 5 and 12 years

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 590 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Participants' physical activity will be measure over the course of 5 consecutive school days pre-intervention and 5 consecutive school days post-intervention
  Accelerometer and SOPLAY observation

SECONDARY OUTCOMES:
Change in dietary intake | Participants' dietary intake will be measure over the course of 5 consecutive school days pre-intervention and 5 consecutive school days post-intervention
  plate waste consumption

CONTACTS AND LOCATIONS:
Overall Officials: Steven Gortmaker, PhD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard Prevention Research Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Virgara R, Phillips A, Lewis LK, Baldock K, Wolfenden L, Ferguson T, Richardson M, Okely A, Beets M, Maher C. Interventions in outside-school hours childcare settings for promoting physical activity amongst schoolchildren aged 4 to 12 years. Cochrane Database Syst Rev. 2021 Sep 27;9(9):CD013380. doi: 10.1002/14651858.CD013380.pub2. PMID 34694005
- [Derived] Lee RM, Giles CM, Cradock AL, Emmons KM, Okechukwu C, Kenney EL, Thayer J, Gortmaker SL. Impact of the Out-of-School Nutrition and Physical Activity (OSNAP) Group Randomized Controlled Trial on Children's Food, Beverage, and Calorie Consumption among Snacks Served. J Acad Nutr Diet. 2018 Aug;118(8):1425-1437. doi: 10.1016/j.jand.2018.04.011. PMID 30055710
- [Derived] Cradock AL, Barrett JL, Giles CM, Lee RM, Kenney EL, deBlois ME, Thayer JC, Gortmaker SL. Promoting Physical Activity With the Out of School Nutrition and Physical Activity (OSNAP) Initiative: A Cluster-Randomized Controlled Trial. JAMA Pediatr. 2016 Feb;170(2):155-62. doi: 10.1001/jamapediatrics.2015.3406. PMID 26641557
- [Derived] Lee RM, Emmons KM, Okechukwu CA, Barrett JL, Kenney EL, Cradock AL, Giles CM, deBlois ME, Gortmaker SL. Validity of a practitioner-administered observational tool to measure physical activity, nutrition, and screen time in school-age programs. Int J Behav Nutr Phys Act. 2014 Nov 28;11:145. doi: 10.1186/s12966-014-0145-5. PMID 25429898
- [Derived] Giles CM, Kenney EL, Gortmaker SL, Lee RM, Thayer JC, Mont-Ferguson H, Cradock AL. Increasing water availability during afterschool snack: evidence, strategies, and partnerships from a group randomized trial. Am J Prev Med. 2012 Sep;43(3 Suppl 2):S136-42. doi: 10.1016/j.amepre.2012.05.013. PMID 22898163